CLINICAL TRIAL: NCT05130853
Title: Social Cognition Individualized Activities Lab (SoCIAL) for the Training of Social Cognition and Narrative Enhancement in Patients With Schizophrenia: A Randomized Controlled Study to Assess Efficacy and Generalization to Real-life Functioning
Brief Title: Efficacy Study of a New Individualized Rehabilitation Programme for Social Cognition in Patients With Schizophrenia
Acronym: SoCIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Silvana Galderisi, Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4870/2020
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: cognitive remediation; psychiatric rehabilitation; social cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoCIAL Group (Experimental): Subjects will conduct SoCIAL programme once a week, for a total of 10 weeks. Every session consists of two different modules: 1) a training programme that helps patients recognize emotions and important social signals (such as facial expressions and prosody) and develop strategy focused on the Theory of Mind; 2) a training in narrative enhancement. Time of administration for both modules is 30 minutes; the operator, however, can choose to focus the session on one module rather than the other, based on the subject's specific needs.
  Interventions: Behavioral: Social Skills and Neurocognitive Individualized Training (SoCIAL); Other: Treatmment-as-usual
- Control Group - Treatment-as-usual (TAU) (Active Comparator): Subjects that will be randomized in this group will receive their treatment as usual for the whole length of the study (10 weeks). TAU includes all the psychiatric therapies (pharmacological, psychological, occupational etc) that subjects may have begun before study's enrollment.
  Interventions: Other: Treatmment-as-usual

INTERVENTIONS:
Behavioral: Social Skills and Neurocognitive Individualized Training (SoCIAL) — SoCIAL is composed of two modules:
  1. Social Cognition Training The Emotions recognition training will train the subject's ability in discriminating between different emotional states through photos and videos. The Theory of Mind (ToM) training will help subjects discriminate between emotional expressions in social contexts and understand other people's mental state with videos that display actors expressing several emotional states. More details in Palumbo et al., 2017.
  2. Narrative Enhancement Training The narrative enhancement training consists in story-telling exercises focused on improving the subject's capacity to comprehend his/her emotional experience.
  Arms: SoCIAL Group
Other: Treatmment-as-usual — Subjects that will be randomized in this group will receive their treatment as usual for the whole length of the study. TAU includes all the psychiatric therapies (pharmacological, psychological, occupational etc) that subjects may have begun before study's enrollment.

SUMMARY:
Patients affected by schizophrenia often present significant deficits in various aspects of social cognition, such as social perception, recognition of one's own and other people's emotional state and the theory of mind. Recent studies investigated the correlation between social cognition and real-life functioning, reporting that greater social cognition deficits determine worse social and occupational functioning in real-life.

Therefore, social cognition deficits represent an important target both in therapeutic and rehabilitative treatment in patients with psychotic conditions, especially in the early phases of the disease.

Our research group has implemented a new individualized rehabilitation programme for social cognition: the Social Cognition Individualized Activities Lab, SoCIAL. The pivotal study showed that this programme improves specifically social cognition abilities, even when compared to a standardised and validated rehabilitation programme such as the Social Skills And Neurocognitive Individualized Training (SSANIT). However, the improvement in social cognition did not translate in improvement in real-life functioning.

Recently, another key aspect that plays a role in quality of life and real life functioning in people with schizophrenia has emerged, the narrative abilities. Available data confirm that this variable has a strong impact on social functioning and quality of life in patients with schizophrenia.

Taking into account the above evidence, our group decided to implement a new version of the social cognitive remediation programme in order to overcome the limitations found during its pivotal study. The new SoCIAL programme is characterized by specific modules for training of social cognition and narrative abilities in patients with schizophrenia. The efficacy of this programme, compared to treatment as usual, in individuals diagnosed with schizophrenia or schizoaffective disorder will be assessed. The generalization of improvement to real-life functioning domains will also be evaluated in completers and in the intent-to-treat sample.

DETAILED DESCRIPTION:
BACKGROUND:

In patients with schizophrenia an impairment in different cognitive domains has been well established. Cognitive impairment has been associated with poor social functioning and poor quality of life. Evidence has been reported suggesting that the impact of cognitive impairment in real-life functioning is even greater than the one exerted by positive and negative symptoms. Furthermore, this impairment can be detected throughout different phases of schizophrenia, such as the premorbid, prodromal and remission stages of the illness. From a neurobiological perspective, this impairment might be explained as the cumulative effect of abnormalities in neuronal maturation processes, neurodevelopment and neuroplasticity that could lead to defective cortico-cerebellar-thalamic-cortical circuits.

Among all the cognitive domains, Social Cognition (SC) was highlighted not only for its direct impact on functioning, but also for its key role in mediating the effects of the other cognitive domains on real-life functioning. SC represents a complex cognitive domain that underlies fundamental abilities for social interactions, such as the capacity to perceive, interpret and generate answers based on other people's intentions, emotions, and behaviors.

Studies regarding SC in schizophrenia identified 4 sub-domains impaired in affected subjects: emotion recognition, social role perception, theory of mind and attributional style.

Despite the key role that cognitive impairment plays in schizophrenia, the pharmacological options of treatment against them seem to have a marginal impact; consequently, a number of psychological treatments has been developed in order to get a significant improvement in the cognitive domains impairments, in quality of life and in real-life functioning. Specifically, the cognitive remediations programmes are mainly targeted in improving neurocognitive functions (such as attention, memory, learning) rather than obtaining a better outcome in SC, even if the early results in this field are promising.

Different approaches have been used to develop cognitive remediation programmes for SC: some of them, defined as "integrated", aim to train both SC domains and neurocognitive domains; other programmes, defined as "targeted", are designed to improve only specific SC domains. A meta-analysis of SC programmes showed that these interventions produce significant improvements in 2 of the 4 SC impaired domains in schizophrenia (facial emotion recognition and theory of mind), as well as in real life functioning and in negative symptoms.

The Department of Psychiatry of the University of Campania "Luigi Vanvitelli" developed an integrated group intervention, the Social Cognition Individualized Activities Lab (SoCIAL), with the purpose to improve both SC domains (recognition of emotions and theory of mind). In the pivotal study, SoCIAL was compared to a largely validated remediation programme for social abilities, the Social Skills and Neurocognitive Individualized Training. Results showed that participants that underwent the SoCIAL programme improved their SC abilities, together with a significant reduction of the avolition domain in negative symptomatology, compared to the control group.

Conversely, no difference was found among the two groups when looking at other clinical variables such as positive and disorganized symptoms, neurocognitive functions and real-life functioning. In particular, any of the participants in both groups showed an improvement in social functioning, probably due to the "rooftop effect", i.e. the high level of functioning that these patients already had before the treatment started.

The main limitations found for this programme concerned two aspects: 1) the conduction of the intervention in a group setting and 2) the role-play module. The group setting was considered to be bounding because: a) in a group session, it is harder to individualize the intervention, considering that it could be challenging to work on deficits shared by all participants); b) participants' recruitment could be complicated if some subjects refuse, or are unable, to attend group sessions. The role-play, a very useful technique for the treatment of social abilities, does not seem to have the same results when it comes to SC; the SoCIAL programme, in fact, aims to improve one's capacity to recognize other people's emotions, thoughts and beliefs. During the role-play simulation, subjects may experience frustration in case they are unable to understand the role played by another patient during the simulation, considering that the intentions of the "actor" should be hidden to the subject.

Additionally, literature has recently identified an interesting technique that could help individuals affected by schizophrenia train their narrative ability, i.e. narrative enhancement. A consensual definition of "narrative abilities" is complicated by the multitude of theoretical approaches. According to the phenomenological perspective, narrative abilities consist of two different components: phenomenological continuity and narrative continuity. Phenomenological continuity is the ability to make "mental time travel", both reliving past experiences and pre-experiencing events that may occur in the future. Narrative continuity is the sense of personal continuity due to the ability to create a personal story (biography) that is coherent and adherent to the facts. These abilities are impaired in schizophrenia and several studies have shown a correlation between narrative abilities and metacognition. Narrative and metacognitive abilities play a substantial role in determining the poor quality of life for people with schizophrenia and low personal narrative ability is also associated with negative and depressive symptoms. Some studies used the narrative enhancement technique in a rehabilitation programme defined as "integrated", since it trained both neurocognitive and narrative abilities. The results are encouraging, considering that this technique seems to considerably decrease internalized stigma and to improve quality of life for participants, even when compared to other psychological and rehabilitative programmes.

This project aims to evaluate the efficacy of the SoCIAL programme in a larger sample. Moreover, it will be administered individually (not in a group setting) and the narrative enhancement technique will replace the role-play session (more info available in "Social Cognitive Individualized Activities Lab" paragraph, in "Methods" section). Lastly, the efficacy of the programme will be evaluated by comparing the SoCIAL's participants vs a group of patients treated as usual.

AIMS:

1. to modify and implement the individualized cognitive remediation programme (SOcial Cognition Individualized Activities Lab, SoCIAL)
2. to compare the efficacy of SoCIAL programme vs (treatment-as-usual (TAU) in patients that have been diagnosed with schizophrenia/schizoaffective disorder (based on DSM-V criteria) with illness durations <10 years. Efficacy will be evaluated with primary and secondary outcomes: 1) the primary outcome is to evaluate SoCIAL efficacy on patients' social cognition, negative symptoms, level of functioning and quality of life; 2) the secondary outcome is to evaluate improvements in positive and disorganized symptoms of schizophrenia, functional capacity and cognition.

PROCEDURE:

The study will be carried out at The Department of Psychiatry of the University of Campania "Luigi Vanvitelli" and the Department of Mental Health and Addictions, ASST Fatebenefratelli Sacco that will enroll outclinic patients with a diagnosis of schizophrenia/schizoaffective disorder according to DSM-V criteria, confirmed by Structured Clinical Interview for DSM-5 - Patient version (SCID-I-P) There will be 80 enrolled subjects (40 for each center). Subjects will be randomly assigned to the SoCIAL or the TAU group. Overall, 40 patients (20 for each center) will be assigned to SoCIAL and 40 (20 for each center) to TAU. Subjects will be evaluated before the programme starts and as soon as it ends. Following eligibility and baseline assessment participants are randomly assigned to either an intervention or control (TAU) group using an Excel spreadsheet. The investigators stratified randomisation considering age, gender and years of education.

The study will have a total length of 12 months, divided in these phases:

1) Operators will be trained in evaluating neurocognitive functions, social cognition, functional capacity and real life functioning ; 2) Operators will also be trained in SoCIAL programme's practice; 3) Recruitment of patients and randomization (in both centers); 4) assessment of neurocognitive functions, social cognition, functional capacity and real life functioning for enrolled patients; 5) implementation of interventions; 6) assessment of neurocognitive functions, social cognition, functional capacity and real life functioning in subjects at the end of the programme for both group (SoCIAL programme vs TAU); 7) final evaluation and data analysis.

DATA ANALYSIS:

An assessment of the statistical power of this study was performed by an effect size's analysis of the studies included in a recent meta-analysis (Kurtz and Richardson 2012). The results are very satisfactory: with a statistical power ≥0.8 and a significance level of <.05, our study needs a total sample of 68 subjects as against the 80 subjects that the investigators are recruiting.

Neuropsychological, psychopathological and cognitive functioning evaluations will be conducted pre and post interventions. Statistical analysis will be conducted by ANOVA for repeated measures, focusing on the role played by different types of interventions in each group regarding the aforementioned domains.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia/schizoaffective disorder according to DSM-V criteria, in stabilized phase of the disease;
* Illness duration <10 years;
* No major pharmacological treatment modifications in the last 3 months;
* Minimum 5 years of education.

Exclusion Criteria:

* Organic diseases that cause disabilities;
* Usual consumption of alcohol and drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Positive Symptoms | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  The Positive and Negative Syndrome Scale (PANSS, administration time = 30') will be used for the evaluation of positive symptoms. The PANSS is a semistructured interview composed of 30 items divided in three subscales, namely positive symptoms, negative symptoms, and general psychopathology. Each item is accompanied by a specific definition and by detailed anchoring criteria for each rating point, ranging from "absent" (1) to "severe" (7). According to the five-factor model proposed by Wallwork et al. (2012), the investigators will calculate the positive dimension by summing the scores on the items "Delusions" (P1), "Hallucinatory behavior" (P3), "Grandiosity" (P5) and "Unusual thought content (G9).
Negative Symptoms | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  The Positive and Negative Syndrome Scale (PANSS, administration time = 30') will be used for the evaluation of positive symptoms. The PANSS is a semistructured interview composed of 30 items divided in three subscales, namely positive symptoms, negative symptoms, and general psychopathology. Each item is accompanied by a specific definition and by detailed anchoring criteria for each rating point, ranging from "absent" (1) to "severe" (7). According to the five-factor model proposed by Wallwork et al. (2012), the investigators will calculate the negative dimension by summing the scores on the items "Blunted Affect" (N1), "Emotional Withdrawal" (N2), "Poor Rapport" (N3), "Passive/Apathetic Social Withdrawal" (N4) and "Lack of spontaneity" (N6).
Disorganization | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  The Positive and Negative Syndrome Scale (PANSS, administration time = 30') will be used for the evaluation of the disorganized symptoms. The PANSS is a semistructured interview composed of 30 items divided in three subscales, namely positive symptoms, negative symptoms, and general psychopathology. Each item is accompanied by a specific definition and by detailed anchoring criteria for each rating point, ranging from "absent" (1) to "severe" (7). According to the five-factor model proposed by Wallwork et al. (2012), the disorganization dimension will be calculated with three PANSS items: "Conceptual disorganization" (P2), "Difficulty in abstract thinking" (N5), and "Poor attention" (G11).
Neurocognitive functions | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  Neurocognitive functions will be assessed using the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB). This test includes items designed to evaluate six neurocognitive domains: a) processing speed; b) attention and vigilance; c) working memory; d) verbal learning and memory; e) visual learning and memory; f) reasoning and problem solving (administration time = 80').
  9 tests are included to measure neurocognitive domains (Category Fluency - Animal Naming; Brief Assessment of Cognition in Schizophrenia Symbol Coding; Trail Making Test - Part A; Continuous Performance Test - Identical Pairs; Wechsler Memory Scale Spatial Span; Letter-Number Span; Hopkins Verbal Learning Test - Revised; Brief Visuospatial Memory Test - Revised; Neuropsychological Assessment Battery - Mazes).
Social cognition | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  Social cognition will be evaluated with the Mayer-Salovey-Caruso Emotional Intelligence Test included in the MCCB battery.
  To better assess social cognition (in addition to the MSCEIT) participants will undergo the Facial Emotional Identification Test (FEIT, administration time = 15') as well as the The Awareness of Social Inference Test (TASIT, evaluation time = 15'), a theory of the mind measure. The FEIT involves black-and-white photographs of 19 different individuals' faces (nine females/10 males) each depicting one of six different emotions (happiness, sadness, anger, surprise, fear, shame), shown one at a time for 15 s. After each stimulus, the participant should select which of the six emotions better describe the picture shown. The Awareness of Social Inference Test (TASIT) is a measure of basic emotion perception and complex social cognition. This test evaluates social cognition through videotaped vignettes designed to reflect the real life interactions.
General cognitive abilities | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  General cognitive abilities will be evaluated with the Wechsler Adult Intelligence Scale-Revised (WAIS-R). This instrument is a revised form of the WAIS, a test that consisted of six verbal and five performance subtests. The WAIS-R uses four subtests (arithmetic, block design, picture completion, and information) to estimate verbal and performance IQ that are highly correlated with the full WAIS assessments.
Functional ability | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  Functional ability will be assessed by the brief version of UCSD Performance-based Skills Assessment (UPSA-Brief, administration time = 15'), an instrument that measures participants' capacity to perform tasks similar to those encountered in daily life. The UPSA-B consists of two of the five subscales from the full UPSA: 1) Financial skills and 2) Communication skills. For the assessment of financial skills, participants are given fake money to handle (for example, they are asked to count them, make change, pay bills). Assessment of communication skills involves tasks in which participants use a disconnected landline telephone to simulate phone calls (e.g., doctor's office) to communicate requested or necessary information. The final score (calculated by summing the two subscales scores) ranges from 0 to 100, with higher scores indicating better functional capacity.
Functioning | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  The Specific Level of Functioning Scale (SLOF, administration time = 20') will be used to evaluate the subject's functioning. This scale consists of 43 items and relies on data reported by an operator and on the direct observation of subejct's behaviors and functioning in several domains: (1) physical functioning, (2) personal care skills, (3) interpersonal relationships, (4) social acceptability, (5) activities of community living and (6) work skills.
Quality of Life assessment | Pre (T0) and Post (T1) Intervention - 3 Months time frame
  Quality of life will be measured through the Quality of Life Scale (QOLS, administration time = 5'), a semi-structured interview, composed by 21 items, designed to assess four different areas of psychosocial adjustment, including Interpersonal Relations, Instrumental Role (e.g., work, school, homemaker), Intrapsychic Foundations (e.g., motivation, sense of purpose), and Common Objects and Activities (e.g., owning a watch, use of public transportation).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maj, MD, PhD, Study Director — Department of Psychiatry - University of Campania "Luigi Vanvitelli"
Locations (1):
- Department of Psychiatry - University of Campania "Luigi Vanvitelli", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galderisi S, Bucci P, Mucci A, Kirkpatrick B, Pini S, Rossi A, Vita A, Maj M. Categorical and dimensional approaches to negative symptoms of schizophrenia: focus on long-term stability and functional outcome. Schizophr Res. 2013 Jun;147(1):157-162. doi: 10.1016/j.schres.2013.03.020. Epub 2013 Apr 19. PMID 23608244
- [Background] Galderisi S, Davidson M, Kahn RS, Mucci A, Boter H, Gheorghe MD, Rybakowski JK, Libiger J, Dollfus S, Lopez-Ibor JJ, Peuskens J, Hranov LG, Fleischhacker WW; EUFEST group. Correlates of cognitive impairment in first episode schizophrenia: the EUFEST study. Schizophr Res. 2009 Dec;115(2-3):104-14. doi: 10.1016/j.schres.2009.09.022. Epub 2009 Oct 12. PMID 19822407
- [Background] Galderisi S, Maj M, Mucci A, Cassano GB, Invernizzi G, Rossi A, Vita A, Dell'Osso L, Daneluzzo E, Pini S. Historical, psychopathological, neurological, and neuropsychological aspects of deficit schizophrenia: a multicenter study. Am J Psychiatry. 2002 Jun;159(6):983-90. doi: 10.1176/appi.ajp.159.6.983. PMID 12042187
- [Background] Green MF, Harvey PD. Cognition in schizophrenia: Past, present, and future. Schizophr Res Cogn. 2014 Mar;1(1):e1-e9. doi: 10.1016/j.scog.2014.02.001. PMID 25254156
- [Background] Green MF, Kern RS, Braff DL, Mintz J. Neurocognitive deficits and functional outcome in schizophrenia: are we measuring the "right stuff"? Schizophr Bull. 2000;26(1):119-36. doi: 10.1093/oxfordjournals.schbul.a033430. PMID 10755673
- [Background] Galderisi S, Rucci P, Mucci A, Rossi A, Rocca P, Bertolino A, Aguglia E, Amore M, Bellomo A, Bozzatello P, Bucci P, Carpiniello B, Collantoni E, Cuomo A, Dell'Osso L, Di Fabio F, di Giannantonio M, Gibertoni D, Giordano GM, Marchesi C, Monteleone P, Oldani L, Pompili M, Roncone R, Rossi R, Siracusano A, Vita A, Zeppegno P, Maj M; Italian Network for Research on Psychoses. The interplay among psychopathology, personal resources, context-related factors and real-life functioning in schizophrenia: stability in relationships after 4 years and differences in network structure between recovered and non-recovered patients. World Psychiatry. 2020 Feb;19(1):81-91. doi: 10.1002/wps.20700. PMID 31922687
- [Background] Moritz S, Silverstein SM, Dietrichkeit M, Gallinat J. Neurocognitive deficits in schizophrenia are likely to be less severe and less related to the disorder than previously thought. World Psychiatry. 2020 Jun;19(2):254-255. doi: 10.1002/wps.20759. No abstract available. PMID 32394552
- [Background] Mucci A, Rucci P, Rocca P, Bucci P, Gibertoni D, Merlotti E, Galderisi S, Maj M; Italian Network for Research on Psychoses. The Specific Level of Functioning Scale: construct validity, internal consistency and factor structure in a large Italian sample of people with schizophrenia living in the community. Schizophr Res. 2014 Oct;159(1):144-50. doi: 10.1016/j.schres.2014.07.044. Epub 2014 Aug 30. PMID 25182540
- [Background] Schmidt SJ, Mueller DR, Roder V. Social cognition as a mediator variable between neurocognition and functional outcome in schizophrenia: empirical review and new results by structural equation modeling. Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S41-54. doi: 10.1093/schbul/sbr079. PMID 21860046
- [Background] Karow A, Wittmann L, Schottle D, Schafer I, Lambert M. The assessment of quality of life in clinical practice in patients with schizophrenia. Dialogues Clin Neurosci. 2014 Jun;16(2):185-95. doi: 10.31887/DCNS.2014.16.2/akarow. PMID 25152657
- [Background] Grant PM, Best MW, Beck AT. The meaning of group differences in cognitive test performance. World Psychiatry. 2019 Jun;18(2):163-164. doi: 10.1002/wps.20645. No abstract available. PMID 31059607
- [Background] Galderisi S, Rossi A, Rocca P, Bertolino A, Mucci A, Bucci P, Rucci P, Gibertoni D, Aguglia E, Amore M, Bellomo A, Biondi M, Brugnoli R, Dell'Osso L, De Ronchi D, Di Emidio G, Di Giannantonio M, Fagiolini A, Marchesi C, Monteleone P, Oldani L, Pinna F, Roncone R, Sacchetti E, Santonastaso P, Siracusano A, Vita A, Zeppegno P, Maj M; Italian Network For Research on Psychoses. The influence of illness-related variables, personal resources and context-related factors on real-life functioning of people with schizophrenia. World Psychiatry. 2014 Oct;13(3):275-87. doi: 10.1002/wps.20167. PMID 25273301
- [Background] Velligan DI, Mahurin RK, Diamond PL, Hazleton BC, Eckert SL, Miller AL. The functional significance of symptomatology and cognitive function in schizophrenia. Schizophr Res. 1997 May 3;25(1):21-31. doi: 10.1016/S0920-9964(97)00010-8. PMID 9176924
- [Background] Davidson M. Cognitive impairment as a diagnostic criterion and treatment target in schizophrenia. World Psychiatry. 2019 Jun;18(2):171-172. doi: 10.1002/wps.20651. No abstract available. PMID 31059612
- [Background] Bond GR, Drake RE, Becker DR. An update on Individual Placement and Support. World Psychiatry. 2020 Oct;19(3):390-391. doi: 10.1002/wps.20784. No abstract available. PMID 32931093
- [Background] Melle I. Cognition in schizophrenia: a marker of underlying neurodevelopmental problems? World Psychiatry. 2019 Jun;18(2):164-165. doi: 10.1002/wps.20646. No abstract available. PMID 31059634
- [Background] Reichenberg A, Velthorst E, Davidson M. Cognitive impairment and psychosis in schizophrenia: independent or linked conditions? World Psychiatry. 2019 Jun;18(2):162-163. doi: 10.1002/wps.20644. No abstract available. PMID 31059615
- [Background] Fatouros-Bergman H, Cervenka S, Flyckt L, Edman G, Farde L. Meta-analysis of cognitive performance in drug-naive patients with schizophrenia. Schizophr Res. 2014 Sep;158(1-3):156-62. doi: 10.1016/j.schres.2014.06.034. Epub 2014 Jul 30. PMID 25086658
- [Background] Kotov R, Jonas KG, Carpenter WT, Dretsch MN, Eaton NR, Forbes MK, Forbush KT, Hobbs K, Reininghaus U, Slade T, South SC, Sunderland M, Waszczuk MA, Widiger TA, Wright AGC, Zald DH, Krueger RF, Watson D; HiTOP Utility Workgroup. Validity and utility of Hierarchical Taxonomy of Psychopathology (HiTOP): I. Psychosis superspectrum. World Psychiatry. 2020 Jun;19(2):151-172. doi: 10.1002/wps.20730. PMID 32394571
- [Background] Heckers S, Kendler KS. The evolution of Kraepelin's nosological principles. World Psychiatry. 2020 Oct;19(3):381-388. doi: 10.1002/wps.20774. PMID 32931122
- [Background] Sitskoorn MM, Aleman A, Ebisch SJ, Appels MC, Kahn RS. Cognitive deficits in relatives of patients with schizophrenia: a meta-analysis. Schizophr Res. 2004 Dec 1;71(2-3):285-95. doi: 10.1016/j.schres.2004.03.007. PMID 15474899
- [Background] Mesholam-Gately RI, Giuliano AJ, Goff KP, Faraone SV, Seidman LJ. Neurocognition in first-episode schizophrenia: a meta-analytic review. Neuropsychology. 2009 May;23(3):315-36. doi: 10.1037/a0014708. PMID 19413446
- [Background] Menon V. Brain networks and cognitive impairment in psychiatric disorders. World Psychiatry. 2020 Oct;19(3):309-310. doi: 10.1002/wps.20799. No abstract available. PMID 32931097
- [Background] Reininghaus U, Bohnke JR, Chavez-Baldini U, Gibbons R, Ivleva E, Clementz BA, Pearlson GD, Keshavan MS, Sweeney JA, Tamminga CA. Transdiagnostic dimensions of psychosis in the Bipolar-Schizophrenia Network on Intermediate Phenotypes (B-SNIP). World Psychiatry. 2019 Feb;18(1):67-76. doi: 10.1002/wps.20607. PMID 30600629
- [Background] Tripathi A, Kar SK, Shukla R. Cognitive Deficits in Schizophrenia: Understanding the Biological Correlates and Remediation Strategies. Clin Psychopharmacol Neurosci. 2018 Feb 28;16(1):7-17. doi: 10.9758/cpn.2018.16.1.7. PMID 29397662
- [Background] Gross G, Huber G. [Schizophrenia: neurodevelopmental disorder or degenerative brain process?]. Fortschr Neurol Psychiatr. 2008 May;76 Suppl 1:S57-62. doi: 10.1055/s-2008-1038153. German. PMID 18461546
- [Background] Galderisi S, Rossi A, Rocca P, Bertolino A, Mucci A, Bucci P, Rucci P, Gibertoni D, Aguglia E, Amore M, Blasi G, Comparelli A, Di Giannantonio M, Goracci A, Marchesi C, Monteleone P, Montemagni C, Pinna F, Roncone R, Siracusano A, Stratta P, Torti MC, Vita A, Zeppegno P, Chieffi M, Maj M; Italian Network for Research on Psychoses. Pathways to functional outcome in subjects with schizophrenia living in the community and their unaffected first-degree relatives. Schizophr Res. 2016 Aug;175(1-3):154-160. doi: 10.1016/j.schres.2016.04.043. Epub 2016 May 19. PMID 27209527
- [Background] Barch DM. Nonsocial and social cognitive function in psychosis: interrelationships, specificity and innovative approaches. World Psychiatry. 2019 Jun;18(2):117-118. doi: 10.1002/wps.20653. No abstract available. PMID 31059631
- [Background] Harvey PD, Penn D. Social cognition: the key factor predicting social outcome in people with schizophrenia? Psychiatry (Edgmont). 2010 Feb;7(2):41-4. PMID 20376275
- [Background] Green MF, Leitman DI. Social cognition in schizophrenia. Schizophr Bull. 2008 Jul;34(4):670-2. doi: 10.1093/schbul/sbn045. Epub 2008 May 20. PMID 18495642
- [Background] Green MF, Lee J, Wynn JK. Experimental approaches to social disconnection in the general community: can we learn from schizophrenia research? World Psychiatry. 2020 Jun;19(2):177-178. doi: 10.1002/wps.20734. No abstract available. PMID 32394575
- [Background] Green MF, Horan WP, Lee J. Nonsocial and social cognition in schizophrenia: current evidence and future directions. World Psychiatry. 2019 Jun;18(2):146-161. doi: 10.1002/wps.20624. PMID 31059632
- [Background] Hill SK, Bishop JR, Palumbo D, Sweeney JA. Effect of second-generation antipsychotics on cognition: current issues and future challenges. Expert Rev Neurother. 2010 Jan;10(1):43-57. doi: 10.1586/ern.09.143. PMID 20021320
- [Background] Keefe RSE. Why are there no approved treatments for cognitive impairment in schizophrenia? World Psychiatry. 2019 Jun;18(2):167-168. doi: 10.1002/wps.20648. No abstract available. PMID 31059617
- [Background] Falkai P, Schmitt A. The need to develop personalized interventions to improve cognition in schizophrenia. World Psychiatry. 2019 Jun;18(2):170. doi: 10.1002/wps.20650. No abstract available. PMID 31059619
- [Background] Roe D, Hasson-Ohayon I, Mashiach-Eizenberg M, Derhy O, Lysaker PH, Yanos PT. Narrative enhancement and cognitive therapy (NECT) effectiveness: a quasi-experimental study. J Clin Psychol. 2014 Apr;70(4):303-12. doi: 10.1002/jclp.22050. Epub 2013 Oct 2. PMID 24114797
- [Background] Missel M, Birkelund R. Ricoeur's narrative philosophy: A source of inspiration in critical hermeneutic health research. Nurs Philos. 2020 Apr;21(2):e12254. doi: 10.1111/nup.12254. Epub 2019 May 14. PMID 31087495
- [Background] Raffard S, D'Argembeau A, Lardi C, Bayard S, Boulenger JP, Van der Linden M. Narrative identity in schizophrenia. Conscious Cogn. 2010 Mar;19(1):328-40. doi: 10.1016/j.concog.2009.10.005. Epub 2009 Dec 1. PMID 19955004
- [Background] Kern RS, Nuechterlein KH, Green MF, Baade LE, Fenton WS, Gold JM, Keefe RS, Mesholam-Gately R, Mintz J, Seidman LJ, Stover E, Marder SR. The MATRICS Consensus Cognitive Battery, part 2: co-norming and standardization. Am J Psychiatry. 2008 Feb;165(2):214-20. doi: 10.1176/appi.ajp.2007.07010043. Epub 2008 Jan 2. PMID 18172018
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Moore RC, Paolillo EW, Heaton A, Fazeli PL, Jeste DV, Moore DJ. Clinical utility of the UCSD Performance-Based Skills Assessment-Brief (UPSA-B) in adults living with HIV: Associations with neuropsychological impairment and patient-reported everyday functioning difficulties. PLoS One. 2017 Aug 24;12(8):e0183614. doi: 10.1371/journal.pone.0183614. eCollection 2017. PMID 28837678
- [Background] Kurtz MM, Richardson CL. Social cognitive training for schizophrenia: a meta-analytic investigation of controlled research. Schizophr Bull. 2012 Sep;38(5):1092-104. doi: 10.1093/schbul/sbr036. Epub 2011 Apr 27. PMID 21525166
- [Background] Yanos PT, Lysaker PH, Silverstein SM, Vayshenker B, Gonzales L, West ML, Roe D. A randomized-controlled trial of treatment for self-stigma among persons diagnosed with schizophrenia-spectrum disorders. Soc Psychiatry Psychiatr Epidemiol. 2019 Nov;54(11):1363-1378. doi: 10.1007/s00127-019-01702-0. Epub 2019 Apr 1. PMID 30937510
- [Background] Alle MC, d'Argembeau A, Schneider P, Potheegadoo J, Coutelle R, Danion JM, Berna F. Self-continuity across time in schizophrenia: An exploration of phenomenological and narrative continuity in the past and future. Compr Psychiatry. 2016 Aug;69:53-61. doi: 10.1016/j.comppsych.2016.05.001. Epub 2016 May 6. PMID 27423345
- [Background] Lysaker PH, Buck KD, Taylor AC, Roe D. Associations of metacognition and internalized stigma with quantitative assessments of self-experience in narratives of schizophrenia. Psychiatry Res. 2008 Jan 15;157(1-3):31-8. doi: 10.1016/j.psychres.2007.04.023. Epub 2007 Nov 19. PMID 18023881
- [Background] Lysaker PH, Dimaggio G, Buck KD, Carcione A, Nicolo G. Metacognition within narratives of schizophrenia: associations with multiple domains of neurocognition. Schizophr Res. 2007 Jul;93(1-3):278-87. doi: 10.1016/j.schres.2007.02.016. Epub 2007 Apr 3. PMID 17407806
- [Background] Lysaker PH, Carcione A, Dimaggio G, Johannesen JK, Nicolo G, Procacci M, Semerari A. Metacognition amidst narratives of self and illness in schizophrenia: associations with neurocognition, symptoms, insight and quality of life. Acta Psychiatr Scand. 2005 Jul;112(1):64-71. doi: 10.1111/j.1600-0447.2005.00514.x. PMID 15952947
- [Background] Palumbo D, Mucci A, Piegari G, D'Alise V, Mazza A, Galderisi S. SoCIAL - training cognition in schizophrenia: a pilot study. Neuropsychiatr Dis Treat. 2017 Jul 20;13:1947-1956. doi: 10.2147/NDT.S136732. eCollection 2017. PMID 28790830
- [Background] Davidson M, Galderisi S, Weiser M, Werbeloff N, Fleischhacker WW, Keefe RS, Boter H, Keet IP, Prelipceanu D, Rybakowski JK, Libiger J, Hummer M, Dollfus S, Lopez-Ibor JJ, Hranov LG, Gaebel W, Peuskens J, Lindefors N, Riecher-Rossler A, Kahn RS. Cognitive effects of antipsychotic drugs in first-episode schizophrenia and schizophreniform disorder: a randomized, open-label clinical trial (EUFEST). Am J Psychiatry. 2009 Jun;166(6):675-82. doi: 10.1176/appi.ajp.2008.08060806. Epub 2009 Apr 15. PMID 19369319
- [Background] Sahakian BJ, Savulich G. Innovative methods for improving cognition, motivation and wellbeing in schizophrenia. World Psychiatry. 2019 Jun;18(2):168-170. doi: 10.1002/wps.20649. No abstract available. PMID 31059610
- [Background] Bowie CR. Cognitive remediation for severe mental illness: state of the field and future directions. World Psychiatry. 2019 Oct;18(3):274-275. doi: 10.1002/wps.20660. No abstract available. PMID 31496075
- [Background] McKenna P, Leucht S, Jauhar S, Laws K, Bighelli I. The controversy about cognitive behavioural therapy for schizophrenia. World Psychiatry. 2019 Jun;18(2):235-236. doi: 10.1002/wps.20636. No abstract available. PMID 31059624
- [Background] Vancampfort D, Firth J, Correll CU, Solmi M, Siskind D, De Hert M, Carney R, Koyanagi A, Carvalho AF, Gaughran F, Stubbs B. The impact of pharmacological and non-pharmacological interventions to improve physical health outcomes in people with schizophrenia: a meta-review of meta-analyses of randomized controlled trials. World Psychiatry. 2019 Feb;18(1):53-66. doi: 10.1002/wps.20614. PMID 30600626
- [Background] Glenthoj LB, Mariegaard LS, Fagerlund B, Jepsen JRM, Kristensen TD, Wenneberg C, Krakauer K, Medalia A, Roberts DL, Hjorthoj C, Nordentoft M. Effectiveness of cognitive remediation in the ultra-high risk state for psychosis. World Psychiatry. 2020 Oct;19(3):401-402. doi: 10.1002/wps.20760. No abstract available. PMID 32931108
- [Background] Muth V, Gyure T, Varadi E. [The cognitive paradigm in the rehabilitation of schizophrenia - focusing on cognitive remediation]. Neuropsychopharmacol Hung. 2015 Sep;17(3):129-40. Hungarian. PMID 26485743
- [Background] Lindenmayer JP, McGurk SR, Khan A, Kaushik S, Thanju A, Hoffman L, Valdez G, Wance D, Herrmann E. Improving social cognition in schizophrenia: a pilot intervention combining computerized social cognition training with cognitive remediation. Schizophr Bull. 2013 May;39(3):507-17. doi: 10.1093/schbul/sbs120. Epub 2012 Nov 3. PMID 23125396
- [Background] Penn DL, Roberts DL, Combs D, Sterne A. Best practices: The development of the Social Cognition and Interaction Training program for schizophrenia spectrum disorders. Psychiatr Serv. 2007 Apr;58(4):449-51. doi: 10.1176/ps.2007.58.4.449. PMID 17412842
- [Background] Wolwer W, Frommann N. Social-cognitive remediation in schizophrenia: generalization of effects of the Training of Affect Recognition (TAR). Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S63-70. doi: 10.1093/schbul/sbr071. PMID 21860049
- [Background] Combs DR, Tosheva A, Penn DL, Basso MR, Wanner JL, Laib K. Attentional-shaping as a means to improve emotion perception deficits in schizophrenia. Schizophr Res. 2008 Oct;105(1-3):68-77. doi: 10.1016/j.schres.2008.05.018. Epub 2008 Jun 27. PMID 18585899
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Roberts DL, Penn DL. Social cognition and interaction training (SCIT) for outpatients with schizophrenia: a preliminary study. Psychiatry Res. 2009 Apr 30;166(2-3):141-7. doi: 10.1016/j.psychres.2008.02.007. Epub 2009 Mar 9. PMID 19272654
- [Background] Nijman SA, Veling W, van der Stouwe ECD, Pijnenborg GHM. Social Cognition Training for People With a Psychotic Disorder: A Network Meta-analysis. Schizophr Bull. 2020 Sep 21;46(5):1086-1103. doi: 10.1093/schbul/sbaa023. PMID 32162658
- [Background] Galderisi S, Piegari G, Mucci A, Acerra A, Luciano L, Rabasca AF, Santucci F, Valente A, Volpe M, Mastantuono P, Maj M. Social skills and neurocognitive individualized training in schizophrenia: comparison with structured leisure activities. Eur Arch Psychiatry Clin Neurosci. 2010 Jun;260(4):305-15. doi: 10.1007/s00406-009-0078-1. Epub 2009 Oct 15. PMID 19826855
- [Background] Bucci P, Piegari G, Mucci A, Merlotti E, Chieffi M, De Riso F, De Angelis M, Di Munzio W, Galderisi S. Neurocognitive individualized training versus social skills individualized training: a randomized trial in patients with schizophrenia. Schizophr Res. 2013 Oct;150(1):69-75. doi: 10.1016/j.schres.2013.07.053. Epub 2013 Aug 18. PMID 23962828
- [Background] Ching EYN, Smyth L, De Souza T, Charlesworth G. The Adaptation and Feasibility of Narrative Enhancement and Cognitive Therapy (NECT) for Late-Onset Psychosis. Community Ment Health J. 2020 Feb;56(2):211-221. doi: 10.1007/s10597-019-00495-5. Epub 2019 Oct 29. PMID 31664623
- [Background] Moritz S, Klein JP, Lysaker PH, Mehl S. Metacognitive and cognitive-behavioral interventions for psychosis: new developments . Dialogues Clin Neurosci. 2019 Sep;21(3):309-317. doi: 10.31887/DCNS.2019.21.3/smoritz. PMID 31749655
- [Background] Berna F, Potheegadoo J, Aouadi I, Ricarte JJ, Alle MC, Coutelle R, Boyer L, Cuervo-Lombard CV, Danion JM. A Meta-Analysis of Autobiographical Memory Studies in Schizophrenia Spectrum Disorder. Schizophr Bull. 2016 Jan;42(1):56-66. doi: 10.1093/schbul/sbv099. Epub 2015 Jul 23. PMID 26209548
- [Background] Raffard S, Esposito F, Boulenger JP, Van der Linden M. Impaired ability to imagine future pleasant events is associated with apathy in schizophrenia. Psychiatry Res. 2013 Oct 30;209(3):393-400. doi: 10.1016/j.psychres.2013.04.016. Epub 2013 May 8. PMID 23664297
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Mucci A, Vignapiano A, Bitter I, Austin SF, Delouche C, Dollfus S, Erfurth A, Fleischhacker WW, Giordano GM, Gladyshev I, Glenthoj B, Gutter K, Hofer A, Hubenak J, Kaiser S, Libiger J, Melle I, Nielsen MO, Papsuev O, Rybakowski JK, Sachs G, Ucok A, Wojciak P, Galderisi S. A large European, multicenter, multinational validation study of the Brief Negative Symptom Scale. Eur Neuropsychopharmacol. 2019 Aug;29(8):947-959. doi: 10.1016/j.euroneuro.2019.05.006. Epub 2019 Jun 27. PMID 31255394
- [Background] Peralta V, Cuesta MJ. Psychometric properties of the positive and negative syndrome scale (PANSS) in schizophrenia. Psychiatry Res. 1994 Jul;53(1):31-40. doi: 10.1016/0165-1781(94)90093-0. PMID 7991730
- [Background] Liang S, Yu W, Ma X, Luo S, Zhang J, Sun X, Luo X, Zhang Y. Psychometric properties of the MATRICS Consensus Cognitive Battery (MCCB) in Chinese patients with major depressive disorder. J Affect Disord. 2020 Mar 15;265:132-138. doi: 10.1016/j.jad.2020.01.052. Epub 2020 Jan 14. PMID 32090734
- [Background] Boone DE. Evaluation of Kaufman's short forms of the WAIS-R with psychiatric inpatients. J Clin Psychol. 1992 Mar;48(2):239-45. doi: 10.1002/1097-4679(199203)48:23.0.co;2-6. PMID 1573027
- [Background] Erol A, Mete L, Sonmez I, Unal EK. Facial emotion recognition in patients with schizophrenia and their siblings. Nord J Psychiatry. 2010;64(1):63-7. doi: 10.3109/08039480903511399. PMID 20092378
- [Background] McDonald S, Bornhofen C, Shum D, Long E, Saunders C, Neulinger K. Reliability and validity of The Awareness of Social Inference Test (TASIT): a clinical test of social perception. Disabil Rehabil. 2006 Dec 30;28(24):1529-42. doi: 10.1080/09638280600646185. PMID 17178616
- [Background] McDonald S, Flanagan S, Rollins J, Kinch J. TASIT: A new clinical tool for assessing social perception after traumatic brain injury. J Head Trauma Rehabil. 2003 May-Jun;18(3):219-38. doi: 10.1097/00001199-200305000-00001. PMID 12802165
- [Background] Mausbach BT, Harvey PD, Goldman SR, Jeste DV, Patterson TL. Development of a brief scale of everyday functioning in persons with serious mental illness. Schizophr Bull. 2007 Nov;33(6):1364-72. doi: 10.1093/schbul/sbm014. Epub 2007 Mar 6. PMID 17341468
- [Background] Patterson TL, Goldman S, McKibbin CL, Hughs T, Jeste DV. UCSD Performance-Based Skills Assessment: development of a new measure of everyday functioning for severely mentally ill adults. Schizophr Bull. 2001;27(2):235-45. doi: 10.1093/oxfordjournals.schbul.a006870. PMID 11354591
- [Background] Burckhardt CS, Anderson KL. The Quality of Life Scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. 2003 Oct 23;1:60. doi: 10.1186/1477-7525-1-60. PMID 14613562
- [Background] Sass LA, Parnas J. Schizophrenia, consciousness, and the self. Schizophr Bull. 2003;29(3):427-44. doi: 10.1093/oxfordjournals.schbul.a007017. PMID 14609238
- [Background] Roe D, Yamin A. [Narrative enhancement and cognitive therapy: A group intervention to reduce self-stigma in people with severe mental illness]. Vertex. 2017 Sep;28(135):384-390. Spanish. PMID 29522586
- [Background] Hansson L, Lexen A, Holmen J. The effectiveness of narrative enhancement and cognitive therapy: a randomized controlled study of a self-stigma intervention. Soc Psychiatry Psychiatr Epidemiol. 2017 Nov;52(11):1415-1423. doi: 10.1007/s00127-017-1385-x. Epub 2017 Apr 19. PMID 28424854
- [Background] Reed GM, First MB, Kogan CS, Hyman SE, Gureje O, Gaebel W, Maj M, Stein DJ, Maercker A, Tyrer P, Claudino A, Garralda E, Salvador-Carulla L, Ray R, Saunders JB, Dua T, Poznyak V, Medina-Mora ME, Pike KM, Ayuso-Mateos JL, Kanba S, Keeley JW, Khoury B, Krasnov VN, Kulygina M, Lovell AM, de Jesus Mari J, Maruta T, Matsumoto C, Rebello TJ, Roberts MC, Robles R, Sharan P, Zhao M, Jablensky A, Udomratn P, Rahimi-Movaghar A, Rydelius PA, Bahrer-Kohler S, Watts AD, Saxena S. Innovations and changes in the ICD-11 classification of mental, behavioural and neurodevelopmental disorders. World Psychiatry. 2019 Feb;18(1):3-19. doi: 10.1002/wps.20611. PMID 30600616
- [Background] Gaebel W, Falkai P, Hasan A. The revised German evidence- and consensus-based schizophrenia guideline. World Psychiatry. 2020 Feb;19(1):117-119. doi: 10.1002/wps.20706. No abstract available. PMID 31922675
- [Background] Harvey PD, Strassnig MT. Cognition and disability in schizophrenia: cognition-related skills deficits and decision-making challenges add to morbidity. World Psychiatry. 2019 Jun;18(2):165-167. doi: 10.1002/wps.20647. No abstract available. PMID 31059625
- [Background] Hasson-Ohayon I, Avidan-Msika M, Mashiach-Eizenberg M, Kravetz S, Rozencwaig S, Shalev H, Lysaker PH. Metacognitive and social cognition approaches to understanding the impact of schizophrenia on social quality of life. Schizophr Res. 2015 Feb;161(2-3):386-91. doi: 10.1016/j.schres.2014.11.008. Epub 2014 Dec 8. PMID 25499045
- [Background] Wallwork RS, Fortgang R, Hashimoto R, Weinberger DR, Dickinson D. Searching for a consensus five-factor model of the Positive and Negative Syndrome Scale for schizophrenia. Schizophr Res. 2012 May;137(1-3):246-50. doi: 10.1016/j.schres.2012.01.031. Epub 2012 Feb 21. PMID 22356801
- [Derived] Giuliani L, Pezzella P, Mucci A, Palumbo D, Caporusso E, Piegari G, Giordano GM, Blasio P, Mencacci C, Torriero S, Galderisi S. Effectiveness of a social cognition remediation intervention for patients with schizophrenia: a randomized-controlled study. Ann Gen Psychiatry. 2024 Dec 28;23(1):52. doi: 10.1186/s12991-024-00535-9. PMID 39732701